CLINICAL TRIAL: NCT02364661
Title: The Influence of Short-term Starvation on Disease Severity and Viral Replication Among Hepatitis B Virus Patients
Brief Title: The Influence of Short-term Starvation on Hepatitis B Virus Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, AMIR SHLOMAI, Dr, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0601-14-RMC
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Starvation; Infection
Keywords: Hepatitis B virus; Metabolovirus
MeSH Terms: conditions — Starvation; Infections; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatitis B virus infected patients (Experimental): HBV patients with detectable viremia will be analyzed for their level of viremia following an over-night starvation (fasting) versus fed state
  Interventions: Behavioral: Over night starvation (fasting)

INTERVENTIONS:
Behavioral: Over night starvation (fasting) — HBV viral load will be analyzed after over-night starvation versus following a morning meal

SUMMARY:
Hepatitis B virus is a small DNA virus that affects 400 million people worldwide. The virus infects the liver and previous studies, done in tissue culture and in animals, have shown that viral replication is affected by metabolic changes occurring in the liver. Specifically, starvation induces HBV gene expression and replication, in parallel to the activation of the gluconeogenesis response, and feeding attenuates viral activity. In this study we are going to recruit HBV patients with detectable viremia and analyze their viral load after an over night starvation versus after a morning meal. Our hypothesis is that following an over-night starvation viral load will be higher than that in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis B virus patients with detectable viremia
* >18 years old
* signed a consent form

Exclusion Criteria:

* patients with malignancy
* Patients with diabetes mellitus
* Alcohol consumption of more than 140grams a week
* Advanced liver disease
* HCV or HIV infection
* Pregnancy
* Mental retardation or unable to understand basic explanation about the study -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
A change in the levels of hepatitis B viremia (HBV viral load) between starvation and fed states | Following an over-night (8-12hours) starvation versus following a morning meal. 6 visits overall, one visit every 2 weeks (12 weeks over all).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shlomai, MD/PhD, Principal Investigator — Rabin Medical Center, Beilinson hospital

REFERENCES:
- [Background] Shlomai A, Paran N, Shaul Y. PGC-1alpha controls hepatitis B virus through nutritional signals. Proc Natl Acad Sci U S A. 2006 Oct 24;103(43):16003-8. doi: 10.1073/pnas.0607837103. Epub 2006 Oct 16. PMID 17043229
- [Background] Shlomai A, Shaul Y. The "metabolovirus" model of hepatitis B virus suggests nutritional therapy as an effective anti-viral weapon. Med Hypotheses. 2008;71(1):53-7. doi: 10.1016/j.mehy.2007.08.032. Epub 2008 Mar 10. PMID 18334285